CLINICAL TRIAL: NCT02405494
Title: Effect of Liquid Volume and the Amount of Incorporated Gas Into a Carbohydrate/Protein Beverage on Satiety: a Response-surface-model Study
Brief Title: Effect of Liquid Volume and the Amount of Incorporated Gas Into a Carbohydrate/Protein Beverage on Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 10029V
Record Dates: First submitted 2015-03-12; First posted 2015-04-01 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Satiety; Appetite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Beverage 1 (Other): Liquid foam consisting of 37 ml liquid with 73% overrun (total volume 65 ml).
  Interventions: Dietary Supplement: Beverage 1
- Beverage 2 (Other): Liquid foam consisting of 37 ml liquid with 427% overrun (total volume 197 ml).
  Interventions: Dietary Supplement: Beverage 2
- Beverage 3 (Other): Liquid foam consisting of 98 ml liquid with 73% overrun (total volume 169 ml).
  Interventions: Dietary Supplement: Beverage 3
- Beverage 4 (Other): Liquid foam consisting of 98 ml liquid with 427% overrun (total volume 514 ml).
  Interventions: Dietary Supplement: Beverage 4
- Beverage 5 (Other): Liquid foam consisting of 25 ml liquid with 250% overrun (total volume 88 ml).
  Interventions: Dietary Supplement: Beverage 5
- Beverage 6 (Other): Liquid foam consisting of 110 ml liquid with 250% overrun (total volume 385 ml).
  Interventions: Dietary Supplement: Beverage 6
- Beverage 7 (Other): 68 ml beverage consisting of 68 ml liquid with 0% overrun (total volume 68 ml).
  Interventions: Dietary Supplement: Beverage 7
- Beverage 8 (Other): Liquid foam consisting of 68 ml liquid with 500% overrun (total volume 405 ml).
  Interventions: Dietary Supplement: Beverage 8
- Beverage 9 (Other): Liquid foam consisting of 68 ml liquid with 250% overrun (total volume 236 ml).
  Interventions: Dietary Supplement: Beverage 9

INTERVENTIONS:
Dietary Supplement: Beverage 1
  Arms: Beverage 1
Dietary Supplement: Beverage 2
  Arms: Beverage 2
Dietary Supplement: Beverage 3
  Arms: Beverage 3
Dietary Supplement: Beverage 4
  Arms: Beverage 4
Dietary Supplement: Beverage 5
  Arms: Beverage 5
Dietary Supplement: Beverage 6
  Arms: Beverage 6
Dietary Supplement: Beverage 7
  Arms: Beverage 7
Dietary Supplement: Beverage 8
  Arms: Beverage 8
Dietary Supplement: Beverage 9
  Arms: Beverage 9

SUMMARY:
Liquid foams can be formed by trapping pockets of gas in a beverage. The primary objective of this study is to test the individual contribution, and possible interaction, of the liquid volume and gas to liquid volume ratio (i.e. %overrun (%OR, defined as 100 x [gas volume/liquid volume]) of a beverage to its satiating properties.

DETAILED DESCRIPTION:
It is not known how the liquid and gas volumes of a liquid foam contribute to its satiating properties and how and if these factors interact. The best way to assess these parameter combinations and their interactions is to use a special statistical approach named "Response Surface Methodology" (RSM). The current study therefore has a Central Composite Design with 9 foams differing in liquid volume and in ratio of gas to liquid volume (%overrun, which is defined as 100 x gas volume/liquid volume).

Each subject will be appointed to a single parameter combination and receives this parameter combination twice, separated by a one-week wash-out period.

On both test days subjects' self-assessment of feelings of satiety and physical discomfort will be recorded during 4 hours post-consumption of the treatment using Electronic Visual Analogue Scale.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 21 and 32 kg/m²
* Apparently healthy: measured by questionnaire: no reported current or previous metabolic diseases or chronic gastrointestinal disorders
* Reported dietary habits: no medically prescribed diet, no slimming diet, used to eat 3 meals a day, no vegetarian.
* Reported intense sporting activities below 10h/w
* Reported alcohol consumption below 14 units/w (female volunteers) or below 21 units/w (male volunteers)

Exclusion Criteria:

* Dislike, allergy or intolerance to test products or indicating to be unable to consume 514 ml of aerated test product
* Any food allergy, or dislike or intolerance with the foods supplied during the study
* Eating disorder (measured by SCOFF questionnaire, 2 or more"yes" responses) High or very high restrained eaters (measured by questionnaire; score of 15 or higher, Polivy et al. 1978)
* Reported medical treatment that may affect eating habits/satiety
* Reported lactating (or lactating < 6 weeks ago), pregnant (or pregnant < 6 months ago) or wish to become pregnant during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2011-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Hunger and satiety questions (Area under the time curve of hunger and satiety scores (as rated by the subjects on a Visual Analog Scale) | 245 minutes
  Area under the time curve of hunger and satiety scores (as rated by the subjects on a Visual Analog Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Leatherhead Food Research, Leatherhead, Surrey, United Kingdom